CLINICAL TRIAL: NCT04102657
Title: Blood Glucose Differences Between Left Arm and Right Arm Using a Continuous Glucose
Brief Title: Blood Glucose Differences Between Left Arm and Right Arm Using a Continuous Glucose Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-04
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Diabetes
Keywords: CGM; Glucose Monitoring; Intermittent Fasting; Fasting; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Intermittent Fasting; Fasting; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Intermittent Fasting with Left Arm Exercise (Experimental): Healthy volunteers willing to fast for a 16-hour period daily for 12-14 days. Volunteers will also complete a 20-minute unilateral arm exercise daily.
  Interventions: Other: Intermittent Fasting; Other: Left Arm Exercise
- Intermittent Fasting with Right Arm Exercise (Experimental): Healthy volunteers willing to fast for a 16-hour period daily for 12-14 days. Volunteers will also complete a 20-minute unilateral arm exercise daily.
  Interventions: Other: Intermittent Fasting; Other: Right Arm Exercise
- Free-living Diet with Left Arm Exercise (Experimental): Healthy volunteers maintaining their current diet for 12-14 days. Volunteers will also complete a 20-minute unilateral arm exercise daily.
  Interventions: Other: Free-Living Diet; Other: Left Arm Exercise
- Free-living Diet with Right Arm Exercise (Experimental): Healthy volunteers maintaining their current diet for 12-14 days. Volunteers will also complete a 20-minute unilateral arm exercise daily.
  Interventions: Other: Free-Living Diet; Other: Right Arm Exercise

INTERVENTIONS:
Other: Intermittent Fasting — Participants will be instructed to limit their daily food consumption to an 8-hour period in the day of their choosing. For the 16-hour fasting period, subjects are to eliminate caloric intake.
  Arms: Intermittent Fasting with Left Arm Exercise; Intermittent Fasting with Right Arm Exercise
Other: Free-Living Diet — Participants will maintain their current daily food consumption with no caloric restriction. Patient must not have participated in a specialized diet or weight loss program within 2 weeks of enrollment.
  Arms: Free-living Diet with Left Arm Exercise; Free-living Diet with Right Arm Exercise
Other: Left Arm Exercise — Participants will complete a 20-minute period of rest followed by a 20-minute unilateral arm exercise on the left arm. In the middle of the study, participants will switch to the right arm to complete their unilateral arm exercises.
  Arms: Free-living Diet with Left Arm Exercise; Intermittent Fasting with Left Arm Exercise
Other: Right Arm Exercise — Participants will complete a 20-minute period of rest followed by a 20-minute unilateral arm exercise on the right arm. In the middle of the study, participants will switch to the left arm to complete their unilateral arm exercises.
  Arms: Free-living Diet with Right Arm Exercise; Intermittent Fasting with Right Arm Exercise

SUMMARY:
Interest in continuous glucose monitors (CGMs) is growing for use in evaluating real time glucose levels and in detecting extreme high and low values. A CGM is a small device primarily placed on the patient's upper arm or abdomen to measure glucose at frequent time intervals. While the accuracy of these devices is researched extensively, there are no large-scale studies evaluating the differences in the right and left arm in terms of device placement. In addition, intermittent fasting has gained popularity due to potential health benefits including reductions in weight, cholesterol, and blood glucose. However, there remains a shortage of studies researching the effect of short-term intermittent fasting on body fat.

The purpose of this study is to see if there is a difference between glucose levels in the right arm and left arm and to examine if short-term intermittent fasting may impact an individual's body fat percentage.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) is an emerging field for diabetes management. CGM allows providers to individualize therapy by looking at real time glucose levels, detect changes in blood glucose and raise awareness for hypo- and hyperglycemic events.[1] Some CGM devices can be placed on the patient's arm to monitor blood glucose every few minutes. The data is then sent to a monitor for visualization. There are multiple Food and Drug Administration (FDA)- approved devices for continuous glucose monitoring. The FDA considers a device to be accurate if 99% of blood glucose measurements are within 20% of lab results and if 95% of blood glucose measurements are within 15% of lab results.[2]

The accuracy and precision of CGM devices is improving with several products gaining FDA approval. CGM data has been deemed accurate for self-use to adjusted insulin dosage, detection of hypoglycemia and determining the clinical response to therapy. However, events of low glucose readings and false alarms have been reported.[3]

An analysis conducted of the reports to the FDA Manufacturer and User Facility Device Experience (MAUDE) database since 2015 revealed over 25,000 complaints of CGM device inaccuracy.[4] Although CGM devices are researched extensively, there are no studies confirming that the measurements amongst the right arm and left arm are the same.

Intermittent fasting is an eating pattern in which individuals alternate between a period (~16 or more hours) of eliminated or restricted food intake, and a period of normal food intake. It has gained popularity in the public due to proposed health benefits including reductions in weight, cholesterol, and blood glucose.[6] There is published evidence that suggests beneficial effects of intermittent fasting on body fat. In an 8-week study, a significant decrease in fat mass was observed in the intermittent fasting group compared to the free-living group (-16.4 vs -2.8%).[8] However, this is the only human study assessing time-restrictive intermittent fasting and its effects on body fat, and there remains a shortage of high-quality evidence. We would like to further expand existing research by assessing the effect of short-term intermittent fasting on body fat.

This study is a controlled, prospective trial that aims to evaluate the difference in glucose readings between the right arm and left arm using continuous glucose monitors. In addition this study aims to evaluate the difference in percent body fat between short-term intermittent fasting and a free-living diet. Subjects will follow their designated diet for 12-14 days. The study will assess any changes in glucose levels, body fat percent, body mass index (BMI), weight, body composition before and after this 12-14 day study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Willing to wear CGM device for 12-14 days on both arms
* Have active health insurance
* Willing to refrain from any heat therapy for the duration of the study
* Having an interest to comply with the fasting requirements of the study as appropriate
* Willingness to maintain once daily email responses

Exclusion Criteria:

* Any active dermatologic condition on the upper arms
* Implanted medical devices (i.e. pacemaker)
* Critically ill or dialysis patients
* Planned magnetic resonance imaging screening, computed tomography scan, x-ray imaging or high-frequency electrical heat treatment during study period
* Current systemic infections
* Subjects who are unable to fully understand the study or consent process will not be included in the study due to the lack of a qualified medical translator
* Refusal to sign the informed consent document
* Pregnant, planned-pregnancy in the next 30 days, or breast-feeding
* Active eating disorder
* Taking any medications that have an increased risk of hypoglycemia (e.g. sulfonylureas, insulin, thiazolidinediones) as determined by the primary investigators
* Taking medications for obesity
* You have one of the following medical conditions that can cause rapid weight loss: rheumatoid arthritis, hyperthyroidism, irritable bowel syndrome, cancer, HIV, active tuberculosis, Addison's disease
* In an active weight loss program
* On a specialized diet (e.g. Weight Watchers, ketogenic diet, Atkins diet)
* Completed a specialized diet in the past 2 weeks (e.g. Weight Watchers, ketogenic diet, Atkins diet)
* History of adverse events (i.e. shaking, dizziness, fatigue, fainting) during any prior fasting experience
* Below the age of 18 years and above the age of 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Difference in time-matched glucose levels between the right arm and left arm | 12-14 days
Difference in body-fat percentage before and after 12-14 days of designated diet | 12-14 days

SECONDARY OUTCOMES:
Difference in glucose readings between the right arm and left arm before and after 20-minutes of unilateral arm exercise | 12-14 days
Difference in glucose readings between the right arm and left arm per designated diet | 12-14 days
Change in Body Mass Index before and after 12-14 days of designated diet | 12-14 days
Change in Body Fat Analysis before and after 12-14 days of designated diet | 12-14 days
Difference in percent of total glucose readings in hypoglycemic range (Interstitial BG <70mg/dL) between the right arm and left arm | 12-14 days
Difference in percent of total glucose readings in euglycemic range (Interstitial BG 70mg/dL-180mg/dL) between the right arm and left arm | 12-14 days
Difference in percent of total glucose readings in hyperglycemic range (Interstitial BG >180mg/dL) between the right arm and left arm | 12-14 days
Difference in percent of total glucose readings in hypoglycemic range (Interstitial BG <70mg/dL) between designated diet groups | 12-14 days
Difference in percent of total glucose readings in euglycemic range (Interstitial BG 70mg/dL-180mg/dL) between designated diet groups | 12-14 days
Difference in percent of total glucose readings in hyperglycemic range (Interstitial BG >180mg/dL) between designated diet groups | 12-14 days
Time in range (Interstitial BG 70mg/dL-180mg/dL) between the right arm and left arm | 12-14 days
Time below range (Interstitial BG <70 mg/dL) between the right arm and left arm | 12-14 days
Time in range (Interstitial BG 70mg/dL-180mg/dL) between designated diet groups | 12-14 days
Time below range (Interstitial BG <70 mg/dL) between designated diet groups | 12-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Pacific, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2. Food and Drug Administration. Self-monitoring blood glucose test systems for over-the-counter use-guidance for industry and food and drug administration staff. Available at: http://www.fda.gov/downloads/MedicalDevices/DeviceRegulationandGuidance/GuidanceDocuments/UCM380327.pdf. Accessed October 10, 2016.
- [Background] 1. Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group, Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D: The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care 2009;32:1378-1383
- [Background] Rodbard D. Continuous Glucose Monitoring: A Review of Successes, Challenges, and Opportunities. Diabetes Technol Ther. 2016 Feb;18 Suppl 2(Suppl 2):S3-S13. doi: 10.1089/dia.2015.0417. PMID 26784127
- [Background] Shapiro AR. Nonadjunctive Use of Continuous Glucose Monitors for Insulin Dosing: Is It Safe? J Diabetes Sci Technol. 2017 Jul;11(4):833-838. doi: 10.1177/1932296816688303. Epub 2017 Mar 1. PMID 28540756
- [Background] Stote KS, Baer DJ, Spears K, Paul DR, Harris GK, Rumpler WV, Strycula P, Najjar SS, Ferrucci L, Ingram DK, Longo DL, Mattson MP. A controlled trial of reduced meal frequency without caloric restriction in healthy, normal-weight, middle-aged adults. Am J Clin Nutr. 2007 Apr;85(4):981-8. doi: 10.1093/ajcn/85.4.981. PMID 17413096
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Derived] Kawakatsu S, Liu X, Tran B, Tran BP, Manzanero L, Shih E, Shek A, Lim JJ. Differences in Glucose Readings Between Right Arm and Left Arm Using a Continuous Glucose Monitor. J Diabetes Sci Technol. 2022 Sep;16(5):1183-1189. doi: 10.1177/19322968211008838. Epub 2021 May 6. PMID 33955249